CLINICAL TRIAL: NCT07352072
Title: Incidence of Bleeding, Thrombosis and Transfusion Requirements in ICU Patients With COVID-19 Supported With Veno-venous Extracorporeal Membrane Oxygenation: a Single-center Retrospective Cohort Study
Brief Title: Incidence of Bleeding, Thrombosis and Transfusion Requirements in ICU Patients With COVID-19 Supported With Veno-venous Extracorporeal Membrane Oxygenation
Status: Not yet recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Vibeke Lind Jørgensen, MD, pHD, consultant, Rigshospitalet, Denmark
Other Study IDs: P-2025-19510; R-25054929 (Other: team for journaldata)
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: VV ECMO; Bleeding; Thrombosis; Transfusion Adverse Reaction; COVID-19
MeSH Terms: conditions — Hemorrhage; Thrombosis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with COVID-19 induced ARDS supported with VV ECMO in eastern Denmark: a single-center retrospective cohort study of all adult ICU patients with COVID-19 infection supported with veno-venous extracorporeal membrane oxygenation admitted to the cardio-thoracic intensive care unit at Copenhagen University Hospital, Rigshospitalet.

SUMMARY:
The investigators aim to assess the risk of bleeding and thrombo-embolic complications as well as benefit and harm of blood product transfusion and anticoagulation therapy in adult ICU patients with COVID-19 supported with V-V ECMO

DETAILED DESCRIPTION:
During the SARS-CoV-2 (COVID-19) pandemic millions of people were affected worldwide, some only experiencing minor symptoms whilst some developed acute respiratory distress syndrome (ARDS) requiring admission to the intensive care unit (ICU). ARDS is a life-threatening condition with mortality ranging from 35-48 %. Gas exchange can be severely impaired and, in some cases, conventional mechanical ventilation and adjunct therapies cannot accomplish adequate oxygenation. Veno-venous extracorporeal membrane oxygenation (V-V ECMO) is recommended as a rescue-support for refractory hypoxemia in ARDS also following COVID-19 infection and has been utilised widely. However, optimal management is difficult with prolonged ECMO duration in ARDS patients with COVID-19 and reported survival rates vary considerably 34-66

%. Complications include severe bleeding requiring more red cell transfusions and thrombotic complications, which are common despite increased risk of bleeding. Both bleeding and thrombosis are associated with increased mortality and balancing the opposing risks is challenging in daily management. On one hand, patients are routinely exposed to anticoagulant therapy (e.g. systemic heparin for the ECMO circuit operation), but on the other hand, patients are commonly exposed to blood product transfusions. The timing, monitoring, efficacy and safety of both blood product transfusion and anticoagulant therapy remains poorly understood. The investigators therefore aim to assess the risk of bleeding and thrombo-embolic complications as well as benefit and harm of blood product transfusion and anticoagulation therapy in adult ICU patients with COVID-19 supported with V-V ECMO.

Objectives

1. To assess the incidence, site and risks of bleeding and thrombo-embolic events in ICU patients with COVID-19 supported with V-V ECMO.
2. To assess the quantity of transfused blood products.
3. To assess the clinical practice of anticoagulant therapy in this cohort.
4. To assess the incidence of transfusions-related serious adverse events.

ELIGIBILITY:
Inclusion criteria:

* Adults
* Polymerase chain reaction (PCR) verified COVID-19 infection
* Supported with V-V ECMO in this center

Exclusion criteria:

- none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators will conduct a single-center retrospective cohort study of all adult ICU patients with COVID-19 infection supported with veno-venous extracorporeal membrane oxygenation admitted to the cardio-thoracic intensive care unit at Copenhagen University Hospital, Rigshospitalet.
  The department represents one of two ECMO sites in Denmark and has a referral area inhabiting approximately 2.75 million people.
  Study period: February 26th 2020 (date of the first officially verified Danish patient infected with COVID-19) until December 31st 2021 (date of the last verified COVID-19 patient supported with V-V ECMO in this center). Patients will be followed from time of specialised ICU admission to death or a maximum of 90 days.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Bleeding events | 90 days
  A bleeding event is defined as any event requiring at least 3 units of red blood cells within 24 hours or transfusion with 3 or more units of either fresh frozen plasma, platelet concentrates or red blood cells within 24 hours, any intracranial bleeding or bleeding requiring invasive/surgical interventions

SECONDARY OUTCOMES:
Thrombo-embolic events | 90 days
  A thrombo-embolic event is defined as any radiologically proven event (i.e. ultrasound, CT- or MRI scan) or any event that led to a significant change in patient management (i.e. changes in anticoagulant therapy or requiring invasive interventions).
Use of blood products transfusion in the ICU | 90 days
  Number of units and estimated volume of red blood cells, platelets, fresh frozen plasma, fibrinogen concentrates, cryoprecipitate and anti-thrombin-III substitution
Use of anticoagulant therapy | 90 days
  Number of days on anticoagulant therapy and type of anticoagulant used in the ICU
Transfusion-related serious adverse events | 90 days
  A serious adverse event defined as any event requiring immediate discontinuation of transfusion or deterioration of any organ system that has previously been unaffected by the underlying disease following transfusion (e.g. anaphylaxis, haemolytic reactions, TRALI, TACO).30

CONTACTS AND LOCATIONS:
Locations (1):
- Department of cardiothoracic anaesthsia and intensive care 4141, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
We dont know if other groups are interested in the data